CLINICAL TRIAL: NCT05060029
Title: A Pilot Study to Evaluate the Efficacy and Safety of Lactobacillus Species Suppositories on Vaginal Health and pH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP/210503/VB/VDPH
Record Dates: First submitted 2021-09-15; First posted 2021-09-28 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-01

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Coconut Oil

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: In order to preserve the blinding, IP and placebo suppositories will be matched for size, shape, color, and texture. They will be packed in identical fashion in terms of size, color, as well as labelling. The blinding will be done at the CRO (Vedic Lifesciences Pvt. Ltd.). The participant IDs will be arranged in chronological order as per the randomization chart. This chart will be secured, saved and maintained in the electronic Trial Master File (TMF) under the respective project folder.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lactobacillus Species Suppositories (Experimental): Coconut oil fatty acids, hyaluronic acid, patented VagiBIOM Probiotic complex CFU (Lactobacillus crispatus Bi16, Lactobacillus gasseri Bi19, Bacillus coagulans Bi34, Lactobacillus acidophilus Bi14) hydrolyzed cellulose, oligofructose, silica gel, lactic acid
  Interventions: Drug: Lactobacillus Species
- Coconut Oil Suppositories (Placebo Comparator): Coconut oil fatty acid suppositories
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lactobacillus Species — Lactobacilli containing suppositories have been successfully used in the past to maintain the vaginal environment and for treatment of infections like BV. Some of the Lactobacilli species that have been used include Lactobacillus acidophilus, Lactobacillus crispatus, Lactobacillus gasseri and Lactobacillus plantarum, none of which demonstrated any safety concerns. The investigational product, which contains a Lactobacilli complex as its main component, has already been marketed as a tool to maintain vaginal microbial balance, pH and the prevention of microbial infection, thus there are no additional safety concerns or risks involved in this clinical trial design.
  Arms: Lactobacillus Species Suppositories
Other: Placebo — Coconut Oil Fatty Acids
  Other Names: Coconut Oil
  Arms: Coconut Oil Suppositories

SUMMARY:
Most of the methods involved in the treatment of BV include antibiotics. Some of the antibiotics used for this include metronidazole, clindamycin and fluconazole. The antibiotics inhibit the growth of anaerobes that support G. vaginalis and other microbes without affecting lactobacilli. This leads to the treatment of BV while also preventing its recurrence. However, the use of antibiotics may lead to antibiotic resistance and cause various side-effects such as thrush, dizziness, rash, nausea, etc. In the case of many antibiotics, the cure rates were incredibly poor and the BV recurrence rates reached as high as 80 %. Probiotic therapy has slowly been replacing antibiotics for the treatment and prevention of BV and other infections. These probiotics usually contain lactobacilli and help maintain a healthy vaginal environment. They can either be consumed through curd and other milk products that contain probiotics (mostly lactobacilli) or they can be used in the form of suppositories that are placed in the vagina. In probiotics containing lactobacilli, the lactic acid produced by the bacteria lowers the vaginal pH to the ideal range of 3.5 to 4.5 and prevents infection recurrence. Lactobacilli containing suppositories have been successfully used in the past to treat BV, being marketed as a safe and effective way to prevent and treat infections for women in various stages of their lives.

DETAILED DESCRIPTION:
The vaginal microbiome is said to be the first line of defence against vaginal infection, due to competitive exclusion and the destruction of pathogenic microbes. The vagina remains relatively sterile until a woman reaches puberty, after which the hormonal changes cause the colonization of lactobacilli in the vaginal environment. Any alterations in the microbiota are seen to cause symptomatic conditions. These conditions may include bacterial vaginosis (BV), vaginal candidiasis and trichomoniasis. The reduction in circulating hormone levels in older women as they near menopause triggers various physiological changes in the vagina. Vulvovaginal atrophy, dryness, itchiness, redness, loss of elasticity, inflammation and atypical secretions are some of the changes that occur in the vagina as estrogen and progesterone levels decrease in the blood.

The aforementioned reduction in hormone levels would also lead to a decline in the concentration of lactobacilli in the vaginal environment. The lactobacilli produce lactic acid, which creates an acidic vaginal environment conducive to the growth of lactobacilli, while preventing the growth of other anaerobic bacterial species. The dominant lactobacilli also prevent the binding of other bacteria to the epithelial cells and the lactic acid produced by lactobacilli blocks histone deacetylases, thereby enhancing gene transcription and DNA repair within their cells. Moreover, the lactobacilli also inhibit the induction of pro-inflammatory cytokines while promoting homeostasis. Some of the species from the Lactobacilli genus that have been identified as residents of the vaginal environment include L. crispatus, L. gasseri, L. iners, and L. jensenii Therefore, it is seen that women who experience lowering of hormone levels i.e. as they approach menopause, the chances of contracting vaginal infection increases due to the lower concentrations of lactobacilli. Bacteria such as Gardnerella, Atopobium, Mobiluncus, Prevotella, Streptococcus, Ureaplasma and Megasphaera, which were previously left dormant due to the lactobacilli, may increase in concentration and increase the susceptibility of these women to contract infections such as bacterial vaginosis.

Bacterial vaginosis is usually caused by the overabundance of G. vaginalis and other anaerobes, and can be clinically diagnosed using the Amsel criteria. This technique requires at least three positive findings of the four diagnostic criteria: a fishy odor after a 10% potassium hydroxide test for vaginal secretion, the presence of non-inflammatory vaginal discharge, clue cells on microscopic examination, and vaginal fluid pH > 4.5. The nugent score is also a well-validated technique to diagnose BV.

In this study, the safety and efficacy of the vaginal suppository VagiBIOM will be studied in aging women with BV infection. The effect of the suppository on vaginal pH and the physiological changes in the vagina will be examined, along with its impact on vaginal infection.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant, non-breastfeeding females between the ages of 40 and 65 years, inclusive.
2. Participants having at least 3 out of following symptoms or signs:

   1. Homogeneous, thin, white discharge that smoothly coats the vaginal walls.
   2. Presence of the clue cells on microscopic examination (as assessed by wet mount test)
   3. pH of vaginal fluid ≥5
   4. A fishy odor of vaginal discharge.
3. Participants with Nugent score of ≥ 7.
4. Participants with a total Vaginal Health Index (VHI) score <15.
5. Participants with pH ≥ 5.
6. Willing to abstain from sexual intercourse 48 hours prior to scheduled clinic visit.
7. Participants able to comply with and perform the procedures requested by the protocol (including IP compliance, blood sample collection procedures and study visit schedule).
8. Participants who are literate enough to understand the essence of study, are informed about the purpose of the study, and understand their rights.
9. Participants able to give written informed consent and willingness to participate in the study and comply with its procedures.

Exclusion Criteria:

1. Participants with signs or symptoms of vaginal or cervical or pelvic or urinary infection on screening or clinical diagnosis of vaginal/cervical/pelvic/ urinary infection in the past 14 days (including but not limited to yeast vulvovaginitis, chlamydia, gonorrhea, trichomonas, genital ulcer disease, pelvic inflammatory disease).
2. Participants who are undergoing Hormone Replacement Therapy (HRT).
3. Participants on prebiotics or probiotics in the last 1 month.
4. Participants who are currently using antibiotics.
5. Participants with history/ signs of cervical or vaginal high grade squamous intraepithelial dysplasia (HSIL), atypical glandular cells of uncertain significance (AGUS) or cervical intraepithelial neoplasia.
6. Participants who have undergone total hysterectomy or any other surgery involving the female reproductive system.
7. Participants who have been diagnosed with polycystic ovary syndrome (PCOS).
8. Uncontrolled type II diabetes mellitus (assessed by RBS ≥140 mg/dL.)
9. Use of an immunosuppressive or immunomodulatory drug within 6 months prior to enrolment.
10. Participants with uncontrolled hypertension defined as systolic blood pressure (SBP) ≥ 140 mm Hg and/or diastolic blood pressure (DBP) ≥ 90 mm Hg).
11. Abnormal Thyroid Stimulating Hormone (TSH) value out of reference range of 0.35 to 5.00 μIU/mL.
12. History of any significant neurological and psychiatric condition which may affect the participation and inference of the study's end points.
13. Participation in other clinical trials in last 3 months prior to screening.
14. Smokers (Past smokers can be allowed if they have abstinence for minimum 2 years).
15. Chronic or sporadic abdominal pain including moderate to severe dysmenorrhoea.
16. Substance abuse problems (within 2 years) defined as:

    1. Use of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.)/Nicotine dependence.
    2. High-risk drinking as defined by consumption of 4 or more alcohol containing beverages on any day or 8 or more alcohol containing beverages per week for women.
17. Any of the following clinically significant illness, i.e. Cardiovascular, endocrine system, immune system, respiratory system, hepatobiliary system, kidney and urinary system, neuropsychiatric, musculoskeletal, inflammatory, blood and tumors, gastrointestinal diseases, etc.
18. History of hepatitis B/ hepatitis C/ HIV infection.
19. Regular medical treatment including over the counter medication, which may have impact on the study aims (e.g., probiotics, antibiotic drugs, laxatives etc.)
20. Any condition that could, in the opinion of the investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-08-12 (Estimated); Study Completion 2022-08-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of IP on Vaginal pH | Day 0 to Day 28
  To evaluate the efficacy of Investigational product (IP) on Vaginal pH as assessed by a pH indicator from baseline to Day 28 in comparison to placebo.

SECONDARY OUTCOMES:
Evaluate the efficacy of IP on Vaginal pH | Day 7 and Day 21
  Vaginal pH as assessed by a pH indicator from baseline to Day 7 and Day 21 in comparison to placebo.
Evaluate the efficacy of IP on Vaginal Itching | Day 0, Day 7, Day 21 and Day 28
  Vaginal itching as assessed by Visual Analogue Scale (0-10) from baseline to Day 28 in comparison to placebo.
Evaluate the efficacy on Microbial Infection control | Day 0, Day 7, Day 21, and Day 28
  Microbial infection control as assessed by the Nugent score from baseline to Day 28 in comparison to placebo.
Evaluate the efficacy as per Vaginal Health Index | Day 0 and Day 28
  Overall Vaginal Health as assessed through clinical examination using the Vaginal Health Index from baseline to Day 28 in comparison to placebo.
Efficacy as per percentage responders in Nugent Score. | Day 0 and Day 28
  Percentage responders as assessed by the number of BV-free women determined using the Nugent score at Day 28 in comparison to placebo.
To evaluate the total number of Adverse Events | Day 7, Day 21, and Day 28
  Number of participants who experienced adverse events from baseline in comparison to placebo

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - JNU Institute for Medical Sciences and Research, Jaipur, Maharashtra
  - Shinde Medicare Hospital, Mumbai, Maharashtra
  - Saraogi Hospital, Mumbai, Maharashtra
  - Shreenika Hospital, Thane, Maharashtra
  - Shubham Sudbhawana Superspeciality Hospital,, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vivekanandan V, Khan ZH, Venugopal G, Musunuru B, Mishra P, Srivastava S, Ramadass B, Subhadra B. VagiBIOM Lactobacillus suppository improves vaginal health index in perimenopausal women with bacterial vaginosis: a randomized control trial. Sci Rep. 2024 Feb 9;14(1):3317. doi: 10.1038/s41598-024-53770-1. PMID 38336815